CLINICAL TRIAL: NCT05001685
Title: Study on the Postoperative Complications and Changes in Posterior Cervical Muscle Volume After Cervical Single Open-door Expansive Laminoplasty With Preservation of Muscular Ligament Complex
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2020161
Record Dates: First submitted 2021-07-01; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-06

CONDITIONS: Cervical Myelopathy
Keywords: Single Open-door Expansive Laminoplasty; Preserving the Unilateral Ligament With Muscle Complex; Postoperative Complications; Effects on Posterior Cervical Muscle Volume
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2006, our hospital improved and began to use cervical expansive open-door laminoplasty preserving the unilateral ligament with muscle complex.The effect of recent follow-up, postoperative complications and their effects on posterior cervical muscle volume were also studied.However, there are few reports about medium and long-term follow-up.

DETAILED DESCRIPTION:
Expansive laminoplasty of posterior cervical canal has been widely used for the treatment of cervical spondylotic myelopathy with cervical spinal stenosis and ossification of the posterior longitudinal ligament since Hirabayashi et al. described it in the 1970s. Traditional single-door surgery requires extensive dissection of both paravertebral muscles and ligaments, and resect part of the spinous process. Postoperative complications (axial neck pain, stiffness, cervical kyphosis, reduced range of motion, etc.) are also related to that in degree. In order to reduce the damage to the posterior cervical structure and reduce the associated complications, in the 1990s, Yoshihiko Oshima et al. introduced the expansive laminoplasty of the spinal canal with one side of the posterior ligamentwith muscle complex attached to the spinous process. In 2006, our hospital improved and began to use cervical expansive open-door laminoplasty preserving the unilateral ligament with muscle complex.The effect of recent follow-up, postoperative complications and their effects on posterior cervical muscle volume were also studied.However, there are few reports about medium and long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* From 2006 to 2018, the patients admitted to the orthopedic department of our hospital for posterior cervical open-door expansive spinal canal laminoplasty with one side muscle-ligament complex reserved.Complete preoperative and postoperative diagnosis and treatment data of our hospital were available, and the follow-up time was ≥2 years.

Exclusion Criteria:

* Patients with incomplete preoperative and postoperative diagnosis and treatment data or less than 2 years of follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From 2006 to 2018, the patients admitted to the orthopedic department of our hospital for posterior cervical open-door expansive spinal canal laminoplasty with one side muscle-ligament complex reserved.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Posterior Cervical Muscle Volume | preoperation
  the volume of Posterior Cervical Muscle
Posterior Cervical Muscle Volume | 2 years after operation
  the volume of Posterior Cervical Muscle
C5 palsy | 2 years after operation
  C5 nerve palsy
axial syndrome | 2 years after operation
  axial syndrome
reoperation | 2 years after operation
  reoperation
door closing | 2 years after operation
  door closing

SECONDARY OUTCOMES:
mJOA | 2 years after operation
  modified Japanese orthopaedics association
NDI | 2 years after operation
  neck disability index
VAS | 2 years after operation
  visual analogue scale
ROM | 2 years after operation
  range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Yu Sun, Dr., Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided